CLINICAL TRIAL: NCT01956916
Title: Effects of LGG Administration in Children With Cystic Fibrosis: A Randomized Controlled Trial
Brief Title: Probiotics in Cystic Fibrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Alfredo Guarino, Full Professor Of Pediatrics, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CF001; 2009-011289-27 (EudraCT Number)
Record Dates: First submitted 2013-09-23; First posted 2013-10-08 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Cystic Fibrosis
Keywords: Pulmonary exacerbation; Inflammation; Intestinal microbiota
MeSH Terms: conditions — Cystic Fibrosis; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotics (Experimental): Capsules containing lyophilized 6x10^9 Colony Forming Units (CFU)/die of Lactobacillus rhamnosus GG (LGG)
  Interventions: Dietary Supplement: Lactobacillus rhamnosus GG
- Placebo (Placebo Comparator): Capsules containing maltodextrin
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus rhamnosus GG — Capsules containing lyophilized 6x10^9 Colony Forming Units (CFU)/die LGG, (60mg) maltodextrin (163 mg), gelatine capsule (75 mg), magnesium stearate (2 mg)
  1 cps/die for 12 months
  Other Names: LGG
  Arms: Probiotics
Dietary Supplement: placebo — Capsules containing maltodextrin (163 mg), gelatine capsule (75 mg), magnesium stearate (2 mg)
  1 cps/die for 12 months
  Arms: Placebo

SUMMARY:
Cystic fibrosis (CF) is a complex systemic disease that mainly involves the respiratory and gastrointestinal (GI) tracts. The polymicrobial community composition of respiratory and GI tracts is influenced by both genetic and environmental factors. Children with CF may harbor an abnormal intestinal microflora, because of altered cystic fibrosis transmembrane conductance regulator (CFTR) function and heavy drug load (antibiotics, pancreatic enzymes and acid suppressors). The investigators have previously demonstrated that intestinal inflammation is highly frequent in CF children, being a major feature of intestinal involvement. In addition, specific probiotics significantly improved airway and GI inflammation in a preliminary trial. The investigators aim to characterize intestinal and respiratory microflora in CF patients and to investigate the effects of daily Lactobacillus GG (LGG) supplementation on both GI and airway microflora and the eventual relationship between probiotic assumption and clinical and inflammation markers. The investigators aim is to eventually improve the quality of life of CF patients, who often suffer from intestinal and respiratory progressive disease, through a non invasive intervention consisting in the supplementation of probiotic bacteria.

ELIGIBILITY:
Inclusion Criteria:

1. A confirmed diagnosis of CF documented by sweat chloride test over 60 mmol/L and confirmed by genotype analysis with the presence of F508del/F508del or F508del/other
2. Boys and girls between 2 and 16 years of age
3. Clinical stability at enrolment, defined as no clinical evidence of acute exacerbation, no modifications in the therapeutic regimen and no hospitalization in the last 2 weeks
4. Pancreatic insufficiency
5. Basal Forced Expiratory Volume 1 second above 50% of predicted value

Exclusion Criteria:

1. Colonization of respiratory tract with Burkholderia cepacia spp.
2. Steroid therapy within one month before enrolment
3. Pregnancy and fertile women taking oral contraceptives
4. Parenteral or oral antibiotics therapy within 2 weeks before enrolment
5. Regular assumption of probiotics
6. Regular assumption of azythromycin

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Actual)
Dates: Start 2010-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in the incidence of pulmonary exacerbations from baseline to 12 months of treatment | every six months up to 18 months
  The incidence of pulmonary exacerbation is assessed every six months. First evaluation from baseline to 6 months of observation. Second evaluation from randomization ( placebo/LGG) to 6 months of treatment and third evaluation after 12 months of treatment
Change of intestinal inflammation from baseline to 12 months of treatment | every six months up to 18 months
  Assessment of intestinal inflammation is performed four times. First time at enrollment, second time at the end of six months of observation. Third time after six months of treatment and fourth time after 12 months of treatment.

SECONDARY OUTCOMES:
Change in the incidence of hospital admission from baseline to 12 months of treatment | every six month up to 18 months
  The incidence of hospital admission is assessed every six months. First evaluation from baseline to 6 months of observation. Second evaluation from randomization ( placebo/LGG) to 6 months of treatment and third evaluation after 12 months of treatment
change in pulmonary function from baseline to 12 months of treatment (measured by Forced Expiratory Volume 1 sec (FEV1)) | every six months up to 18 months
  Assessment of pulmonary function is performed four times. First time at enrollment, second time at the end of six months of observation. Third time after six months of treatment and fourth time after 12 months of treatment.

OTHER OUTCOMES:
Change in the incidence of abdominal pain episodes from baseline to 12 months of treatment | every six months up to 18 months
  The incidence of abdominal pain episodes is assessed every six months. First evaluation from baseline to 6 months of observation. Second evaluation from randomization ( placebo/LGG) to 6 months of treatment and third evaluation after 12 months of treatment
Change in systemic inflammation from baseline to 12 months of treatment | At baseline and after 12 months of treatment
  Assessment of intestinal microflora composition is performed 2 times. First time at randomization (placebo/LGG), second time at the end of 12 months of treatment.
Change of intestinal microflora composition from baseline to 12 months of treatment | baseline and 12 months after treatment
  Assessment of intestinal microflora composition is performed 2 times. First time at randomization (placebo/LGG), second time at the end of 12 months of treatment.

CONTACTS AND LOCATIONS:
Locations (5):
- Italy (5):
  - - Department of Paediatric Medicine, CF Center, "A. Meyer" Children's Hospital, Florence
  - Dipartimento di Pediatria - Università Di Messina, Messina
  - Ospedale Maggiore Policlinico, Mangiagalli e Regina Elena, Milan
  - Università degli studi di Napoli "Federico II", Napoli
  - Ospedale "Bambino Gesù" - Roma, Rome

REFERENCES:
- [Background] Bruzzese E, Raia V, Spagnuolo MI, Volpicelli M, De Marco G, Maiuri L, Guarino A. Effect of Lactobacillus GG supplementation on pulmonary exacerbations in patients with cystic fibrosis: a pilot study. Clin Nutr. 2007 Jun;26(3):322-8. doi: 10.1016/j.clnu.2007.01.004. Epub 2007 Mar 13. PMID 17360077
- [Background] Bruzzese E, Raia V, Gaudiello G, Polito G, Buccigrossi V, Formicola V, Guarino A. Intestinal inflammation is a frequent feature of cystic fibrosis and is reduced by probiotic administration. Aliment Pharmacol Ther. 2004 Oct 1;20(7):813-9. doi: 10.1111/j.1365-2036.2004.02174.x. PMID 15379842
- [Background] Raia V, Maiuri L, de Ritis G, de Vizia B, Vacca L, Conte R, Auricchio S, Londei M. Evidence of chronic inflammation in morphologically normal small intestine of cystic fibrosis patients. Pediatr Res. 2000 Mar;47(3):344-50. doi: 10.1203/00006450-200003000-00010. PMID 10709733
- [Background] Lucidi V, Alghisi F, Raia V, Russo B, Valmarana L, Valmarana R, Coruzzo A, Beschi S, Dester S, Rinaldi D, Maglieri M, Guidotti ML, Ravaioli E, Pesola M, De Alessandri A, Padoan R, Grynzich L, Ratclif L, Repetto T, Ambroni M, Provenzano E, Tozzi AE, Colombo C. Growth assessment of paediatric patients with CF comparing different auxologic indicators: A multicentre Italian study. J Pediatr Gastroenterol Nutr. 2009 Sep;49(3):335-42. doi: 10.1097/MPG.0b013e31818f0a39. PMID 19543116
- [Derived] Miragoli F, Federici S, Ferrari S, Minuti A, Rebecchi A, Bruzzese E, Buccigrossi V, Guarino A, Callegari ML. Impact of cystic fibrosis disease on archaea and bacteria composition of gut microbiota. FEMS Microbiol Ecol. 2017 Feb;93(2):fiw230. doi: 10.1093/femsec/fiw230. Epub 2016 Nov 2. PMID 27810876